CLINICAL TRIAL: NCT01316822
Title: A Study of ARRY-382 in Patients With Selected Advanced or Metastatic Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-382-101
Record Dates: First submitted 2010-12-01; First posted 2011-03-16 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Cancer
Keywords: CSF1R; M-CSF; CSF-1; c-FMS; Tumor-associated macrophage; Macrophage-Colony Stimulating Factor-1; Receptor tyrosine kinase inhibitor; Tumor cell-induced osteolysis
MeSH Terms: conditions — Neoplasm Metastasis

ARMS (1):
- ARRY-382 (Experimental)
  Interventions: Drug: ARRY-382, cFMS inhibitor; oral

INTERVENTIONS:
Drug: ARRY-382, cFMS inhibitor; oral — multiple dose, escalating

SUMMARY:
This is a Phase 1 study during which patients with advanced cancer will receive investigational study drug ARRY-382. Patients will receive increasing doses of study drug in order to achieve the highest dose of the study drug possible that will not cause unacceptable side effects. Patients will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. Approximately 50 patients from the US will be enrolled in this study.

ELIGIBILITY:
Key Inclusion Criteria:

* A histologically or cytologically confirmed diagnosis of advanced or metastatic solid cancer refractory to standard treatment, for which no standard therapy is available or for which the patient refuses standard therapy.
* Measurable disease or evaluable, nonmeasurable disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Hemoglobin ≥ 9.0 g/dL, ANC > 1500/uL and platelet count ≥ 100,000/uL.
* AST/serum glutamic oxaloacetic transaminase (SGOT) and ALT/serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 × the upper limit of normal (ULN).
* Bilirubin ≤ ULN.
* Serum creatinine ≤ 1.5 × ULN.
* Potassium, magnesium and calcium (corrected calcium when serum albumin levels are abnormal) within the normal range.
* Additional criteria exist.

Key Exclusion Criteria:

* 12-lead ECG demonstrating a mean QTcF > 450 msec (triplicate assessment) at the Screening Visit or history/evidence of long QT syndrome.
* History of acute coronary syndromes, including unstable angina, coronary angioplasty, or stenting, within the past 24 weeks.
* Use of concomitant medications that prolong the QT/QTc interval, as assessed by the Investigator, within 14 days prior to first dose of study drug.
* Use of concomitant medication that is a strong CYP3A inhibitor or inducer within 14 days prior to first dose of study drug.
* Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Uncontrolled or symptomatic brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must have been stable for at least 30 days).
* Active refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease) or significant bowel resection that, in the judgment of the Investigator, would preclude adequate absorption (a previous Whipple procedure is allowed).
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the study drug as determined by adverse events, clinical laboratory tests and electrocardiograms. | Safety will be characterized for the duration of time that each patient stays on study; estimated one year.
Establish the maximum tolerated dose (MTD) of study drug. | The MTD will be based on Cycle 1 (28 days).
Characterize the plasma pharmacokinetics (PK) of study drug and its metabolites. | Safety will be characterized for the duration of time that each patient stays on study; estimated one year.

SECONDARY OUTCOMES:
Assess the efficacy of study drug in terms of incidence of response rate and duration of response. | All patients will remain on study until progression of disease, unacceptable toxicity, or another discontinuation criterion is met; estimated one year.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas